CLINICAL TRIAL: NCT04852939
Title: Effectiveness of Bowen's Technique in Patients With Adhesive Capsulitis
Brief Title: Bowen's Technique in Patients With Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00859 Ferwa Tahrim
Record Dates: First submitted 2021-04-20; First posted 2021-04-21 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive capsulitis; Shoulder; Pain; Bowen technique
MeSH Terms: conditions — Bursitis; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bowen's Technique (Experimental): Bowen's Technique
  Interventions: Other: Bowen's technique
- Conventional Physical Therapy (Active Comparator): Conventional Physical Therapy including stretching and strengthening exercises
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Bowen's technique — Initially, cup move is performed which requires a vertically rolling Bowen move over the posterior border of the deltoid muscle above the axillary crease.
  The subject's arm is held flexed at 90 degrees at mid-chest height. Then, the elbow is slowly and passively moved in the direction of the opposite shoulder.
  After maximal adduction of the arm, the therapist firmly taps the lateral aspect of the shoulder with the heel of his/her hand.
  The arm is then carried back to the original start position, where the therapist gently moves superiorly and slightly laterally over the anterior fibers of the deltoid. The arm is then carefully lowered.
  The therapist strives to undertake a minimum of moves and procedures to trigger the body's own self-healing powers and assess how much pressure to use and where and when to perform a move to release the build-up of stress.
  40-minute sessions thrice a week for 6 weeks.
  Arms: Bowen's Technique
Other: Conventional physical therapy — * Hot pack and transcutaneous electrical nerve stimulator (TENS) for 15 minutes.
  * Pendulum stretch, 10 revolutions.
  * Cross body stretch, 4 repetitions.
  * Towel stretch/hand behind the back, 4 repetitions.
  * Isometric internal and external rotation exercises. 40-minute sessions thrice a week for 6 weeks.
  Arms: Conventional Physical Therapy

SUMMARY:
This study will help the physiotherapists in overcoming the challenges and barriers in the treatment. It will also help researchers in acquiring sufficient knowledge for further research on the Bowen technique and its various applications as this technique is not widely applied in the field of physical therapy treatment.

DETAILED DESCRIPTION:
The application of the Bowen technique, producing significant results, will be opted in treatment for the better, improved, and innovative noninvasive management of Adhesive Capsulitis. This study will help the physiotherapists in overcoming the challenges and barriers in the treatment. It will also help researchers in acquiring sufficient knowledge for further research on the Bowen technique and its various applications as this technique is not widely applied in the field of physical therapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age 25 to 60 years
* History of worsening shoulder pain
* Painful movement from at least 3 month
* Grade 2 & 3 adhesive capsulitis
* Both Diabetic and non-diabetic
* Limited Ranges in capsular pattern

Exclusion Criteria:

* Fracture
* Trauma
* Dislocation
* Ongoing physical therapy treatment
* Cortisone injection prior 3 months

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Goniometer | 6th week
  A goniometer is an instrument that either measures an angle or allows an object to be rotated to a precise angular position of joints. Intra-class Correlation Coefficients (ICC≥ 0.94)
Numeric Pain Rating Scale | 6th week
  Numerical Pain Rating Scale (NPRS) the Numerical Rating Scale (NPRS-11) is an 11-points scale for self-report of pain. It is the most commonly used unidimensional pain scale. Interclass correlation coefficient (ICC: 0.74)
Shoulder Pain and Disability Index (SPADI): | 6th week
  self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder. Intra-class correlation coefficient (ICC ≥ 0.89)

CONTACTS AND LOCATIONS:
Overall Officials: Nazish Rafique, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neviaser AS, Neviaser RJ. Adhesive capsulitis of the shoulder. J Am Acad Orthop Surg. 2011 Sep;19(9):536-42. doi: 10.5435/00124635-201109000-00004. PMID 21885699
- [Background] Sathe S, Khurana SK, Damke U, Agrawal PV. To Compare the Effects of Maitland Mobilization with Conventional Physiotherapy in Adhesive Capsulitis. Int J Cur Res Rev| Vol. 2020;12(14).
- [Background] Ewald A. Adhesive capsulitis: a review. Am Fam Physician. 2011 Feb 15;83(4):417-22. PMID 21322517
- [Background] Hand GC, Athanasou NA, Matthews T, Carr AJ. The pathology of frozen shoulder. J Bone Joint Surg Br. 2007 Jul;89(7):928-32. doi: 10.1302/0301-620X.89B7.19097. PMID 17673588
- [Background] Nitsure P, Kothari N. THE EFFECTIVENESS OF BOWEN TECHNIQUE AS AN ADJUNCT TO CONVENTIONAL PHYSIOTHERAPY ON PAIN AND FUNCTIONAL OUTCOMES IN SUBJECT WITH ACUTE TRAPEZITIS-A PILOT STUDY. Romanian Journal of Physical Therapy/Revista Romana de Kinetoterapie. 2015;21(36).
- [Background] Wong PL, Tan HC. A review on frozen shoulder. Singapore Med J. 2010 Sep;51(9):694-7. PMID 20938608
- [Background] Marr M, Baker J, Lambon N, Perry J. The effects of the Bowen technique on hamstring flexibility over time: a randomised controlled trial. J Bodyw Mov Ther. 2011 Jul;15(3):281-90. doi: 10.1016/j.jbmt.2010.07.008. Epub 2010 Sep 15. PMID 21665103
- [Background] Carter B. A pilot study to evaluate the effectiveness of Bowen technique in the management of clients with frozen shoulder. Complement Ther Med. 2001 Dec;9(4):208-15. doi: 10.1054/ctim.2001.0481. PMID 12184347